CLINICAL TRIAL: NCT04439227
Title: MATCH Treatment Subprotocol Z1I: Phase II Study of AZD1775 in Patients With Tumors Containing BRCA1 and BRCA2 Mutations
Brief Title: Testing AZD1775 as a Potential Targeted Treatment in Cancers With BRCA Genetic Changes (MATCH-Subprotocol Z1I)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03212; NCI-2020-03212 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-Z1I (Other: ECOG-ACRIN Cancer Research Group); EAY131-Z1I (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma | interventions — adavosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (adavosertib) (Experimental): Patients receive adavosertib PO QD on days 1-5 and 8-12 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Adavosertib

INTERVENTIONS:
Drug: Adavosertib — Given PO
  Other Names: AZD 1775; AZD-1775; AZD1775; MK 1775; MK-1775; MK1775

SUMMARY:
This phase II MATCH treatment trial identifiesay block the protein tyrosine kinase WEE1 the effects of AZD1775 in patients whose cancer has a genetic change called BRCA mutation. AZD1775 may block a protein called WEE1, which may be needed for growth of cancer cells that express BRCA mutations. Researchers hope to learn if AZD1775 will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive adavosertib (AZD1775) orally (PO) once daily (QD) on days 1-5 and 8-12 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months if less than 2 years from study entry, and then every 6 months for an additional year from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patients must have mutation in the BRCA1 or BRCA2 gene in the tumor, or another aberration, as determined via the MATCH Master Protocol. Patients with tumor carrying mutations defined as variants of uncertain significance will not qualify
* Patients with ovarian cancer or HER2 negative, metastatic breast cancer must have received a PARP inhibitor as part of or as one of their prior lines of therapy
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients receiving any medications or substances that are inhibitors or inducers of CYP3A4, or CYP3A4 substrates need to be reviewed by the study investigator. Continuation of such medications will be at the discretion of the study investigator. Concomitant use of aprepitant and fosaprepitant is prohibited
* Patients have hemoglobin (HgB) >= 9 g/dL, which should be done =< 4 weeks prior to registration to treatment step
* Resting corrected QTc interval using the Fridericia formula (QTcF) should be < 450 msec/male and < 470 msec/female (as calculated per institutional standards) obtained from electrocardiogram (ECG), prior to enrollment. If resting QTc interval using the Fridericia formula (QTcF) is > 450 msec/male and > 470 msec/female (as calculated per institutional standards), then 2 additional ECGs should be performed 2-5 minutes apart at study entry. In order to be eligible, the mean resting corrected QTc interval using the Fridericia formula (QTcF) should be < 450 msec/male and < 470 msec/female (as calculated per institutional standards)

Exclusion Criteria:

* Patients must not have known hypersensitivity to AZD1775 or compounds of similar chemical or biologic composition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-03-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Tumor assessments occurred at baseline, then every 3 cycles until disease progression, up to 3 years post registration
  ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among eligible and treated patients. Objective response rate is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. For each treatment arm, 90% two-sided binomial exact confidence interval will be calculated for ORR.

SECONDARY OUTCOMES:
Overall survival (OS) | Assessed every 3 months for =< 2 years and every 6 months for year 3
  OS is defined as time from treatment start date to date of death from any cause. Patients alive at the time of analysis are censored at last contact date. OS will be evaluated specifically for each drug (or step) using the Kaplan-Meier method.
Progression free survival (PFS) | Assessed at baseline, then every 3 cycles until disease progression, up to 3 years post registration
  Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. PFS will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

DOCUMENTS (1):
  • Study Protocol (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT04439227/Prot_001.pdf